CLINICAL TRIAL: NCT03007940
Title: Using NIATx Strategies to Implement Integrated Services in Routine Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Washington State Department of Social and Health Services (Other); National Institute on Drug Abuse (NIDA) (NIH); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016-0438; R01DA037222 (NIH); 2016-0438 (Other: UW Madison IRB); STUDY00029387 (Other: Study Identifier)
Record Dates: First submitted 2016-12-19; First posted 2017-01-02 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Addiction; Mental Health Disorder
Keywords: Implementation Strategies; Sustainability; Integrated Services
MeSH Terms: conditions — Behavior, Addictive; Mental Disorders | interventions — Commerce

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIATx Strategy (Experimental): The implementation "intervention", NIATx, will be deployed by the first cohort of programs in a 1-year active implementation phase. Each program is assigned an expert quality improvement coach. The coach will help the staff identify ways to improve and integrate services for individuals with co-occurring substance use and mental health disorders. Supports include an in-person coach site visit, coaching including monthly coaching calls and peer to peer coaching calls and learning sessions which promote peer-to-peer sharing about specific goals and objectives and to receive guidance on how to implement organizational level changes to improve integrated treatment services. A walk-through will allow the provider to understand the co-occurring treatment process from a customer perspective.
  Interventions: Other: Coach Site Visit; Other: Walk-through; Other: Learning Sessions; Other: Coaching
- Wait List Control (Placebo Comparator): The wait-list control group will receive the NIATx strategy at the end of the twelve month implementation period for the initial cohort. During the first year of the study, they will follow a business as usual approach to the integration of co-occurring substance use and mental health services.
  Interventions: Other: Business as Usual

INTERVENTIONS:
Other: Coach Site Visit — The coach will conduct a one-day on site visit and will review the walk-through and DDCAT assessment results, and help the change team design an initial change project with Plan-Do-Study-Act (PDSA) cycles. The site visit will use a standardized agenda to ensure NIATx fidelity.
  Arms: NIATx Strategy
Other: Walk-through — Walk-Through: Provider change teams will participate in a coach-led webinar that introduces how to conduct a NIATx walk-through from the co-occurring patient perspective and how to write up results using a standard report format. The walk-through will be conducted within two months of the initial coach site visit.
  Arms: NIATx Strategy
Other: Learning Sessions — The study includes two one-day coach-led learning sessions. The learning sessions promote peer-to-peer sharing about specific goals and objectives. The agenda is tailored to specific treatment service integration issues. The first coach-led learning session teaches providers how to use NIATx process improvement strategies. Providers share walk-through results and initial change projects. Skill development activities include how to: identify change opportunities, use specific tools (e.g., flowcharting), develop PDSA cycles, effectively use data and learning successful change strategies. At the final session, providers present results, sustainment plans, and identify ways for the group to continue to interact.
  Arms: NIATx Strategy
Other: Coaching — A NIATx coach leads the active 12 month implementation phase. The coach works with executive directors, change leaders and teams. After the site visit, a coach will hold individual monthly coaching calls (10 hours in total), and participate in group coaching calls (2 hours in total). In the individual calls, the coach and change team review change projects; discuss successes; and identify ideas for future change projects. Group coaching calls involve change leaders from multiple providers. On these calls, change leaders will discuss common change-related issues, progress, and exchange innovative implementation strategies with their peers. These calls provide opportunities for the coach to share new strategies and discuss implementation issues such as the development of a sustain plan.
  Arms: NIATx Strategy
Other: Business as Usual — Programs in this intervention will continue with their own plans without coaching support to integrate services for individuals with co-occurring substance abuse and mental health disorders. Once the programs in the wait-list control group receive the NIATx Strategy, they will participate in all of the interventions listed above.
  Arms: Wait List Control

SUMMARY:
This is an implementation research study designed to evaluate a defined strategy, NIATx, for its effectiveness in installing and sustaining evidence-based integrated services for persons with co-occurring substance use and mental health disorders. This study is a cluster randomized wait-list control group design, in which a cohort of 25 addiction treatment agencies receives the active NIATx approach during an index 12 month period. The second (wait-list) cohort of 25 addiction treatment agencies activates NIATx strategies during a second index 12 month period. The primary "subjects" of the research are the treatment agencies themselves. The study specific aims are:

1. Relative to wait-list, to determine if NIATx strategies improve implementation outcomes (integrated service fidelity and receipt of more integrated services)
2. Relative to wait-list, to determine if NIATx strategies improve patient care outcomes (psychiatric, alcohol and drug problem severity)
3. Across entire sample, to evaluate variation in the extent of and fidelity to NIATx strategies

NIATx implementation strategies consist of learning sessions, individualized coaching and peer to peer sharing.

ELIGIBILITY:
Inclusion Criteria:

* Organizations who are licensed addiction treatment providers in the state of Washington were identified and provided the opportunity to participate in the study.

Eligibility criteria include:

* outpatient and/or intensive outpatient services
* tax-exempt, government status or at least 50% publicly funded (e.g., block grants, Medicare, Medicaid)
* no prior participation in NIATx research studies (this last criterion excludes 39 agencies who were involved in the NIDA funded NIATx 200)

Exclusion Criteria:

* Public mental health and private addiction treatment agencies are also excluded because only addiction treatment providers in Washington are required to use the state clinical information system, and therefore cannot provide the necessary standardized data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Dual Diagnosis Capability in Addiction Treatment (DDCAT index) scores | Collected at baseline, 12 months, 24 months and 36 months
  DDCAT is a 35-item observational benchmark measure of program level dual diagnosis capability, evaluating policy, clinical practice and workforce dimensions of integrated services for persons with co-occurring disorders.
Change in Penetration Rates: Gain Short Screen | Collected at baseline, 12 months, 24 months and 36 months
  Examine changes in the proportion of program patients screened using the Gain Short Screener. Data for each time point will be collected 90 days before and 90 days after the DDCAT Assessment..
Change in Penetration Rates: Patients receiving integrated medication and psychosocial services | Collected at baseline, 12 months, 24 months and 36 months
  Assessing increased penetration of integrated services based on changes in the proportion of program patients screened, diagnosed and receiving integrated medication and psychosocial services. Data for each time point will be collected 90 days before and 90 days after the DDCAT Assessment.
Change in the Addiction Severity Index (ASI) | Collected at baseline, 12 months, 24 months and 36 months
  Changes in ASI scores for the Psychiatric, Drug and Alcohol composite scores assessed at admission and 30-days post follow-up. Data for each time point will be collected 90 days before and 90 days after the DDCAT Assessment.

OTHER OUTCOMES:
Consolidated Framework for Implementation Research Index | Collected at baseline, 12 months, 24 months and 36 months
  Assess change in Outer Setting, Inner Setting, Characteristics of the Intervention and the Individual Scores as rated by DDCAT Assessor
NIATx Stages of Implementation Completion | Collected during 12 month intervention period
  Assess provider stages of completion related to NIATx intervention based on proportion of activities completed and duration of activities.
NIATx Fidelity | Collected during 12 month intervention period
  Assess fidelity to the NIATx implementation strategies

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ford JH 2nd, Osborne EL, Assefa MT, McIlvaine AM, King AM, Campbell K, McGovern MP. Using NIATx strategies to implement integrated services in routine care: a study protocol. BMC Health Serv Res. 2018 Jun 8;18(1):431. doi: 10.1186/s12913-018-3241-4. PMID 29884164
- [Result] Chokron Garneau H, Assefa MT, Jo B, Ford JH 2nd, Saldana L, McGovern MP. Sustainment of Integrated Care in Addiction Treatment Settings: Primary Outcomes From a Cluster-Randomized Controlled Trial. Psychiatr Serv. 2022 Mar 1;73(3):280-286. doi: 10.1176/appi.ps.202000293. Epub 2021 Aug 4. PMID 34346729
- [Result] Assefa MT, Ford JH 2nd, Osborne E, McIlvaine A, King A, Campbell K, Jo B, McGovern MP. Implementing integrated services in routine behavioral health care: primary outcomes from a cluster randomized controlled trial. BMC Health Serv Res. 2019 Oct 24;19(1):749. doi: 10.1186/s12913-019-4624-x. PMID 31651302
- [Result] Ford JH 2nd, Kaur A, Rao D, Gilson A, Bolt DM, Garneau HC, Saldana L, McGovern MP. Improving Medication Access within Integrated Treatment for Individuals with Co-Occurring Disorders in Substance Use Treatment Agencies. Implement Res Pract. 2021 Jan 1;2:26334895211033659. doi: 10.1177/26334895211033659. Epub 2021 Sep 17. PMID 34988462
- [Derived] Ford JH 2nd, Zehner ME, Schaper H, Saldana L. Adapting the stages of implementation completion to an evidence-based implementation strategy: The development of the NIATx stages of implementation completion. Implement Res Pract. 2023 Sep 19;4:26334895231200379. doi: 10.1177/26334895231200379. eCollection 2023 Jan-Dec. PMID 37790170